CLINICAL TRIAL: NCT00004221
Title: A Phase II Trial Using Multiple Cycles of High Dose Sequential Carboplatin, Paclitaxel and Topotecan With Peripheral Blood Stem Cell (PBSC) Support as Initial Chemotherapy in Patients With Optimally Debulked Stage III Ovarian and Primary Peritoneal Carcinoma
Brief Title: Combination Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Stage III Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9903; NCI-2012-02312 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000067462; GOG-9903 (Other: Gynecologic Oncology Group); GOG-9903 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2000-01-28; First posted 2003-08-25 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Malignant Ovarian Mixed Epithelial Tumor; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Primary Peritoneal Carcinoma; Stage III Ovarian Cancer; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; Paclitaxel; Taxes; Peripheral Blood Stem Cell Transplantation; Topotecan

ARMS (1):
- Treatment (Combination chemotherapy, PBSC) (Experimental): See detailed description.
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Biological: Filgrastim; Drug: Paclitaxel; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Filgrastim — Given SQ
  Other Names: Filgrastim XM02; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo autologous peripheral blood stem cell transplantation
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamptamine; Hycamtin; SKF S-104864-A; Topotecan HCl; topotecan hydrochloride (oral)

SUMMARY:
Phase II trial to study the effectiveness of combination chemotherapy and peripheral stem cell transplantation in treating patients who have undergone surgery for stage III ovarian cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety and feasibility of multiple courses of high dose carboplatin, paclitaxel, and topotecan as initial chemotherapy combined with autologous peripheral blood stem cell transplantation in patients with optimally debulked stage III ovarian or primary peritoneal carcinoma.

II. Determine the pathological complete response rate, disease free survival, and overall survival in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Mobilization and harvest: Within 8 weeks of surgical debulking, patients receive cyclophosphamide IV over 1 hour, followed 4 hours later by paclitaxel IV over 24 hours. Patients receive filgrastim (G-CSF) subcutaneously (SQ) daily beginning 24 hours after completion of paclitaxel infusion and continuing until blood counts recover and autologous peripheral blood stem cells (PBSC) are harvested and selected for CD34+ cells.

High dose chemotherapy and transplantation (3 weeks after PBSC harvest): Patients receive paclitaxel IV over 24 hours beginning on day 1, immediately followed by carboplatin IV over 2 hours, immediately followed by topotecan IV over 24 hours. Patients receive G-CSF sub-cutaneously (SQ) daily beginning 24 hours after completion of topotecan infusion and continuing until blood counts have recovered for 2 days. One quarter of the PBSC are reinfused beginning 2 days after completion of topotecan infusion. Treatment repeats every 4 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with radiographic and biochemical complete response undergo laparoscopy as second look surgery within 8 weeks of the last course of chemotherapy. If no evidence of disease is found during laparoscopy, then exploratory laparotomy must also be performed.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter or at time of recurrence until death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven optimally debulked stage III ovarian or primary peritoneal carcinoma

  * Any of the following subtypes:

    * Serous adenocarcinoma
    * Mucinous adenocarcinoma
    * Clear cell carcinoma
    * Transitional cell carcinoma
    * Endometrioid adenocarcinoma
    * Undifferentiated adenocarcinoma
    * Mixed epithelial adenocarcinoma
    * Adenocarcinoma, not otherwise specified
* No ovarian carcinoma of low malignant potential (borderline)
* Concurrent superficial endometrial or cervical carcinoma allowed if ovarian carcinoma more life threatening or limiting
* Must have undergone appropriate primary surgical staging and debulking for ovarian carcinoma and have less than 1 cm of residual disease

  * No more than 8 weeks since prior surgical debulking
* Must have Hickman catheter in place or be eligible for placement
* No CNS involvement
* Performance status - GOG 0 or 1
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* SGOT or SGPT no greater than 2 times upper limit of normal
* No active hepatitis
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No renal failure
* Curatively treated ureteral obstruction allowed if above creatinine measurements met
* No congestive heart failure
* No myocardial infarction within the past 6 months
* No significant arrhythmias requiring medication
* No poorly controlled systolic or diastolic hypertension (diastolic blood pressure consistently greater than 100 mm Hg)
* No significant nonneoplastic pulmonary disease
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* HIV negative
* No other severe medical or psychiatric illness including, but not limited to the following:

  * Acute infection
  * Active peptic ulcer disease
  * Uncontrolled diabetes mellitus
  * Prior hospitalization for psychiatric illness, including severe depression or psychosis
  * Concurrent alcohol or drug abuse
* No prior chemotherapy for this malignancy
* No radiotherapy to greater than 25% of bone marrow
* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 1999-11; Primary Completion 2002-02-06 (Actual)

PRIMARY OUTCOMES:
Complete response defined as complete disappearance of all measurable and evaluable tumor documented at second-look surgery | Up to 11 years
Indication of excessive toxicity defined as hospitalization > 14 days per course, delay of day 1 therapy > 14 days, or grade 3 (irreversible) or grade 4 vital organ toxicity (non-hematologic) | Up to 11 years

SECONDARY OUTCOMES:
Overall survival | Up to 11 years
PFS | Up to 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schilder, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States